CLINICAL TRIAL: NCT00170781
Title: A 1-Week, Multi-Center, Randomized, Double-Blind, Double-Dummy, Active-Controlled, Parallel Trial Comparing Lumiracoxib (400 mg Once Daily) in Patients With Acute Flares of Gout, Using Indomethacin (50 mg Three Times a Day)
Brief Title: Efficacy and Safety of Lumiracoxib 400 mg Once Daily in Acute Flares of Gout
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2426
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-06

CONDITIONS: Acute Gouty Arthritis
Keywords: Pain, acute gout, arthritis, cyclooxygenase-2 inhibitors, lumiracoxib, indomethacin
MeSH Terms: conditions — Pain; Arthritis | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This study is designed to develop our understanding of the efficacy and safety of using lumiracoxib in the treatment of patients with acute gout. This is a multi-center, double-blind, randomized, parallel group study comparing a single daily dose of 400 mg lumiracoxib with the established dose of indomethacin 50 mg taken three times a day in terms of efficacy

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory cooperative male or female patients of at least 18 years of age
* With an acute attack of gout in 4 joints or less, diagnosed clinically according to the ACR 1977 classification criteria and with an onset within the last 48 hours prior to evaluation. Where more than one joint is involved, the most affected joint should be identified, as the study joint, at baseline and followed throughout the study
* Who present at Baseline with an acute pain intensity of at least moderate.

Exclusion Criteria:

* With an acute attack of gout before the last 48 hours prior to evaluation
* With polyarticular gout involving > 4 joints
* With rheumatoid arthritis, infectious arthritis, pseudo-gout or other acute inflammatory arthritides.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234
Dates: Start 2005-06

PRIMARY OUTCOMES:
Pain intensity in the study joint over days 2 to 5 approximately 4h after the first daily dose

SECONDARY OUTCOMES:
Safety and tolerability profile
Pain intensity in the study joint over the entire treatment period
Patient's and Physician's global assessment of response to therapy
Physician's assessment of tenderness and swelling of study joint
C-reactive protein level
Proportion of patients who discontinued treatment because of a lack of efficacy
Usage of rescue medication
SF-36 and EQ-5D
Physician's assessment of erythema of study joint

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Sponsor GmbH
Locations (2):
- Novartis, Nuremberg, Germany
- For Site Information, contact Novartis Pharma AG, Basel, CH, Switzerland